CLINICAL TRIAL: NCT00197327
Title: Analgesia Requirement and Maternal Satisfaction Following Epidural PCA in Nulliparous Labor: the Effect of a Four-Fold Change in Local Anesthetic Concentration.
Brief Title: Dilute Versus Concentrated Epidural Bupivacaine in Labor
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: Primip-ginosar-HMO-CTIL
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2006-03-03 (Estimated); Status verified 2003-03

CONDITIONS: Pain; Labor Complications
Keywords: Labor Pain; Analgesia, Obstetrical; Pharmacology; Treatment Outcome
MeSH Terms: conditions — Pain; Obstetric Labor Complications; Labor Pain; Agnosia

INTERVENTIONS:
Drug: Epidural bupivacaine (0.25% versus 0.0625%)

SUMMARY:
This study studies labor epidural analgesia and compares dilute (0.0625%) with concentrated (0.25%) bupivacaine.

We hypothesize that patients randomize to receive the concentrated drug will require more drug, will have a more profound motor block, will be more likely to require instrumental delivery and will be less satisfied than those receiving dilute epidural drugs.

DETAILED DESCRIPTION:
This study examines the effect of two different local anesthetic concentrations used for epidural analgesia in labor. Patients are randomized to receive epidural bupivacaine, either as a concentrated (0.25%), or a dilute (0.0625%) solution, both administered by patient-controlled epidural analgesia (PCEA).

ELIGIBILITY:
Inclusion Criteria:

* nulliparity, active spontaneous labor, cervical dilatation greater than 2cm and less than 5 cm, request for epidural analgesia, age between 18 to 40, American Society of Anesthesiologists (ASA) physical status I or II, body weight less than 110kg, gestational age greater than 36 completed weeks, singelton pregnancy and vertex presentation

Exclusion Criteria:

* narcotic administration in the previous 3 hours, non-reassuring fetal heart rate tracing at any stage in labor prior to enrollment, previous uterine surgery, pre-eclampsia and the inability to adequately understand the consent process.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60
Dates: Start 1998-02; Study Completion 2000-03

PRIMARY OUTCOMES:
1. Anesthesia requirement:
a. total dose (mg) of bupivacaine administered
b. number of supplemental bolus doses of bupivacaine self-administered (by PCEA)
c. total number of attempts for supplemental bupivacaine doses (including those denied)

SECONDARY OUTCOMES:
1. Maternal satisfaction (visual analogue scale (VAS) with the anchors being 0 = maximally satisfied and 100 = maximally dissatisfied); after delivery and at 24 hours.
2. Speed of onset of analgesia.
3. Anesthesia variables (in labor q 1hr)
a. Pain score VAS during uterine contraction
b. sensory level
c. motor power
d. maternal blood pressure.
3.Obstetric outcome variables
a. 1st stage duration
b. 2nd stage duration
c. Expulsive efforts
d. Apgar scores at 1 and 5 min
e. Instrumental delivery
f. Cesarean section
g. Non-reassuring fetal heart rate tracing in labor
h. Occipito-posterior malrotation

CONTACTS AND LOCATIONS:
Overall Officials: Yehuda Ginosar, BSc MBBS, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Hebrew University Medical Center, Jerusalem, Israel